CLINICAL TRIAL: NCT04755543
Title: A Phase I Study of Safety and Pharmacokinetics of LP002 (a Humanized Monoclonal Antibody Targeting PD-L1) in Patients With Malignant Digestive System Neoplasms
Brief Title: A Study of LP002 for the Treatment of Patients With Malignant Digestive System Neoplasms
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taizhou HoudeAoke Biomedical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LP002-I-02
Record Dates: First submitted 2021-02-01; First posted 2021-02-16 (Actual); Last update posted 2021-02-16 (Actual); Status verified 2021-02

CONDITIONS: Digestive System Neoplasms
MeSH Terms: conditions — Digestive System Neoplasms | interventions — Cisplatin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- I-A (Experimental): LP002 dose escalation (3+3 design): 6-12 patients with malignant digestive system neoplasms (mainly include gastric/ gastroesophageal junction/ esophageal carcinoma) failed (experienced progressed disease or unable to tolerate) at least one line of previously standard treatment will receive LP002 600mg or 900 mg by intravenous (IV) infusion on Day 1, every 2 weeks (Q2W), for up to 2 year.
  Interventions: Drug: LP002
- I-B (Experimental): If the safety profile in Arm A is acceptable, 9-12 patients with malignant gastric/ gastroesophageal junction carcinoma who are PD-L1 positive and failed (experienced progressed disease or unable to tolerate) at least two lines of previously standard treatments will receive LP002 600mg or 900 mg IV on Day 1, Q2W, for up to 2 year.
  Interventions: Drug: LP002
- I-C (Experimental): If the safety profile in Arm A is acceptable, 15-20 patients with metastatic gastric carcinoma who are PD-L1 positive and systemic treatment-naive will receive LP002 900 mg IV on Day 1, Q2W, and Cisplatin 50mg/m2 IV on Day 1, Q2W, and Fluorouracil 2000 mg/m2 IV continuous infusion over 48 hours from Day 1, Q2W,for up to 2 year.
  Interventions: Drug: LP002; Drug: Cisplatin; Drug: Fluorouracil
- I-D (Experimental): Perioperative treatment: If the safety profile in Arm A is acceptable, 15-20 patients with gastric or gastroesophageal junction carcinoma of cT2-4a, any N, M0 who are PD-L1 positive and systemic treatment-naive will receive LP002 900 mg IV on Day 1, Q2W, and Cisplatin 50mg/m2 IV on Day 1, Q2W, and Fluorouracil 2000 mg/m2 IV continuous infusion over 48 hours from Day 1, Q2W, for 3 cycles, 4-6 weeks before operation of the tumor and receive additional 6 cycles of the same therapy 4 weeks after the operation.
  Interventions: Drug: LP002; Drug: Cisplatin; Drug: Fluorouracil
- I-E (Experimental): Dose escalation (3+3 design) of OH2 (an oncolytic virus) + LP002 900mg：If the safety profile in Arm A is acceptable, 15-30 patients with advanced solid tumors (mainly include digestive system neoplasms) who failed (experienced progressed disease or unable to tolerate) at least one line of previously standard treatment or lack of standard treatments will receive LP002 900mg IV on Day 1, Q2W, and OH2 10^6 or 10^7 or 10^8 CCID50/mL by intra-tumoral injection, Q2W, for up to 2 year.
  Interventions: Drug: LP002; Biological: OH2 oncolytic virus

INTERVENTIONS:
Drug: LP002 — 600mg or 900 mg by intravenous (IV) infusion on Day 1, every 2 weeks (Q2W).
Drug: Cisplatin — 50mg/m2 IV on Day 1, Q2W
  Arms: I-C; I-D
Drug: Fluorouracil — 2000 mg/m2 IV continuous infusion over 48 hours from Day 1, Q2W
  Arms: I-C; I-D
Biological: OH2 oncolytic virus — 106 or 107 or 108 CCID50/mL by intra-tumoral injection, Q2W
  Arms: I-E

SUMMARY:
LP002 is a humanized monoclonal antibody targeting programmed death ligand-1 (PD-L1), which prevents PD-L1 from binding to PD-1 and B7.1 receptors on T cell surface, restores T cell activity, thus enhancing immune response and has potential to treat various types of tumors. In this study, the safety, pharmacokinetics and preliminary efficacy of LP002 for the treatment of malignant digestive system neoplasms will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Understood and signed an informed consent form.
* Age ≥ 18 and ≤ 75 years old, male or female.
* Has histologically confirmed diagnosis of:

Malignant digestive system neoplasms (mainly include gastric/ gastroesophageal junction/ esophageal carcinoma) failed (experienced progressed disease or unable to tolerate) at least one line of previously standard treatment for Arm I-A.

Malignant gastric/ gastroesophageal junction carcinoma who are PD-L1 positive and failed (experienced progressed disease or unable to tolerate) at least two lines of previously standard treatments for Arm I-B.

Metastatic gastric carcinoma who are PD-L1 positive and systemic treatment-naive for Arm I-C.

Gastric or gastroesophageal junction carcinoma of cT2-4a, any N, M0 who are PD-L1 positive and systemic treatment-naive for Arm I-D.

Advanced solid tumors (mainly include digestive system neoplasms) who failed (experienced progressed disease or unable to tolerate) at least one line of previously standard treatment or lack of standard treatments and has suitable lesions for intratumoral injection for Arm I-E.

* Has a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) Performance Score.
* Life expectancy ≥ 3 months.
* Has at least one measurable extracranial lesion according to RECIST1.1 (except Arm-D).
* Has sufficient organ and bone marrow function to meet the following laboratory examination standards:

  1. Blood routine: absolute neutrophil count (ANC)≥1.5×10^9/L; while blood cell count (WBC)≥3×10^9/L; platelet count (PLT)≥100×10^9/L;hemoglobin (HGB)≥90 g/L;
  2. Renal function: Serum creatinine (Scr) ≤1.5×ULN;
  3. Liver function: TBIL≤1.5×ULN; Patients without liver metastases require alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5× ULN. Patients with liver metastases require: ALT and AST≤5×ULN;
  4. The coagulation function is adequate, which is defined as the international normalized ratio (INR) ≤ 2×ULN; or activated partial thromboplastin time (APTT)≤ 1.5×ULN;
* Reproductive men and women of childbearing age are willing to take effective contraceptive measures from signing the informed consent form to 3 months after the last administration of the trial drug.
* Willing to provide tissue samples for PD-L1 biomarker analysis.

Exclusion Criteria:

* Suffered from other malignant tumors in the past 5 years，except those with low risk of metastasis and death (5-year survival rate >90%), for instance, skin basal cell carcinoma, squamous cell carcinoma, and carcinoma in situ from cervix or other regions that have been adequately treated);
* Had prior treatment with any anti-programmed cell death-1 (PD-1), or PD-ligand 1 (PD-L1) or CTLA-4 agent or other immune checkpoint inhibition therapies.
* has active or a history (with high chance of recurrence) of autoimmune diseases, including but not limited to systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, multiple sclerosis, vasculitis, nephritis, except: Type I Diabetes being treated with fixed dose of insulin, hypothyroidism or Hashimoto's thyroiditis that can be controlled only by hormone replacement therapy, skin diseases that do not require systemic treatment (such as eczema, rash covering <10% body surface area, psoriasis without ocular symptoms).
* Expected to undergo major surgery during the study treatment or within 28 days before the first administration of the study drug.
* Has received systemic corticosteroids or other immunosuppressive drugs within 2 weeks before the first administration of the study drug, excluding:

  1. Nasal spray, inhalation or other local glucocorticoids.
  2. Short-term (≤ 7 days) use of glucocorticoids as a preventive medication for allergic reactions or as a therapeutic medication for non-autoimmune diseases.
* Has active digestive ulcer, incomplete intestinal obstruction, active gastrointestinal hemorrhage or perforation.
* Has active interstitial pneumonia, pulmonary fibrosis, acute pulmonary disorders, acute radiation pneumonitis，et al.
* Has uncontrolled systemic diseases, for instance, cardiovascular and cerebrovascular disease, diabetes, tuberculosis.
* Has a history of HIV infection, or other acquired or innate immune deficiency disorders, or a history of organ or stem-cell transplantation.
* Has active chronic HBV or HCV infection, except those with HBV DNA viral load ≤500 IU/mL or <10^3 copies/mL, or HCV RNA negative after adequate treatment.
* Has severe infection within 4 weeks or active infection requiring IV infusion of antibiotics within 2 weeks prior to the first administration of the study drug.
* Known to be allergic to macromolecular protein agents or monoclonal antibody; Known to has a history of severe allergies to any of the components in the study drug;
* Has participated in other clinical trial within 4 weeks before the first administration of the study drug.
* Alcohol dependence or drug abuse within recent one year.
* Has a history of confirmed neurological or mental disorders, such as epilepsy, dementia; or with poor compliance; or the presence of peripheral neurological disorders.
* Has brain metastasis with symptoms.
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial.
* Has received a live vaccine within 30 days prior to the first dose of trial treatment.
* Other reasons disqualifying the entering of this study based on the evaluation of the investigators.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2019-06-17 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | up to approximately 24 months

SECONDARY OUTCOMES:
Objective Response Rate (ORR) for Arm I-A, I-B, I-C, I-E | up to approximately 24 months
  Percentage of subjects achieving complete response (CR) and partial response (PR).
  R0 resection rate RFS pCR
Disease Control Rate (DCR) for Arm I-A, I-B, I-C, I-E | up to approximately 24 months
  Disease Control Rate (DCR) refers to the proportion of subjects who achieve CR, PR and SD through imaging evaluation.
Duration of Response (DOR) for Arm I-A, I-B, I-C, I-E | up to approximately 24 months
  Duration of Response (DOR) is defined as the time from the first evidence of response (PR or CR) to the first evidence of PD or the date of death for any reason.
Progression-Free Survival (PFS) for Arm I-A, I-B, I-C, I-E | up to approximately 24 months
  Progression-free survival (PFS) is defined as the time from the first study drug treatment to disease progression (PD) or to death of the subject due to any reason.
Overall survival (OS) for Arm I-A, I-B, I-C, I-D, I-E | up to approximately 24 months
  Overall survival (OS) refers to the time from the first study drug treatment to death due to any cause.
R0 resection rate for Arm I-D | up to approximately 12 months
  R0 resection rate refers to the rate of patients who have achieved curative resection of the tumor.(Curative resection refers to the absence of tumor after surgical treatment. R0 resection indicates a microscopically margin-negative resection, in which no gross or microscopic tumor remains in the primary tumor bed.)
pathological complete response rate (pCR rate) | up to approximately 12 months
  pathological complete response rate (pCR rate) refers to the rate of patients whose tissue samples show no cancer cells left under a microscope after the anti-cancer treatment.
Terminal half life of LP002 | up to approximately 12 months
Area under curve of LP002 | up to approximately 12 months
Apparent volume of distribution of LP002 | up to approximately 12 months
Systemic clearance of LP002 | up to approximately 12 months
Cmax of LP002 | up to approximately 12 months
Tmax of LP002 | up to approximately 12 months
Serum concentration of the antibody against LP002 within 1 hour prior to each administration | up to approximately 24 months

CONTACTS AND LOCATIONS:
Locations (5):
- China (5):
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Henan Cancer Hospital & Insititute, Zhengzhou, Henan
  - Hubei Cancer Hospital & Insititute, Wuhan, Hubei
  - Liaoning Cancer Hospital & Insititute, Shenyang, Liaoning
  - The First Affiliated Hospital. Zhejiang University School Of Medicine, Hangzhou, Zhejiang